CLINICAL TRIAL: NCT04169555
Title: Impact of the Use of "Point of Care" Ultrasound on the Length of Stay in the Emergency Department During an Episode of Renal Colic
Brief Title: "Point of Care" Ultrasound and Renal Colic
Acronym: ECHOLINE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Lille Catholic University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: RC-P0072
Record Dates: First submitted 2019-11-05; First posted 2019-11-20 (Actual); Last update posted 2019-11-20 (Actual); Status verified 2019-11

CONDITIONS: Renal Colic
Keywords: ultrasound; renal colic; emergency room; point of care
MeSH Terms: conditions — Renal Colic; Emergencies | interventions — High-Energy Shock Waves; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ultrasound (Experimental)
  Interventions: Procedure: Ultrasound
- Standard care (Other)
  Interventions: Other: Standard care

INTERVENTIONS:
Procedure: Ultrasound — The emergency physician will perform a "point of care" ultrasound. If signs of expansions of the pelvicalyceal cavities are found, an early CT scan will follow
  Arms: Ultrasound
Other: Standard care — Standard clinical care of patients. In regards of the clinical evolution and of biological results, a CT scan could be performed by the physician.
  Arms: Standard care

SUMMARY:
The management of renal colic in emergency departments follows the recommendations established at the 8th consensus conference of 2008 on the management of renal colic in emergency services. It recommends the control of pain by nonsteroidal anti-inflammatory drugs and analgesics, the implementation of an urinary test strip and the use of emergency imaging for compiled forms and patient with medical specificities.

Currently, two imaging techniques are recommended during an episode of renal colic:

1. Abdominal x-ray/Ultrasound or non-injected scanner for simple forms to be performed within 24-48h
2. The non-injected scanner for complicated forms In simple forms, the decision to perform any examination remains at the discretion of the physician but with a tendency to carry out a scanner systematically even in the absence of criteria of severity or complication.

The use of the scanner exposes the patient to large doses of radiation even if it is a low dose scanner.

In recent years, studies have been conducted to determine whether the ultrasound, particularly "point of care" ultrasound performed by an emergency physician could be an alternative in the management of renal colic. Studies show that the sensitivity and specificity of ultrasound is comparable to that of the scanner. It has been found that the performance of an ultrasound by the emergency physician allows the decrease in irradiation and also in costs. In 2014,a study published in the New England Journal of Medicine emphasized that the ultrasound performed by the emergency physician would perform just as well as that performed by the radiologist and would result in a decreased time in the emergency room.

The Korean study, published in 2016 in the Clinical and Experimental Emergency Medicine (CEEM), despite some statistical inconsistencies, shows a significant reduction in the time of care by 74 minutes. In this context, we would like to conduct a single-centre, randomised, controlled, open-label study comparing a group of patients benefiting from point of care ultrasound versus a group of patients not benefiting from it. The goal is to determine whether the early ultrasound performed by the emergency physician by detecting expansions of the pelvicalyceal cavities reduces the time spent in the emergency department.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients admitted in ER for suspicion of simple renal colic
* Signed informed consent

Exclusion Criteria:

* protected adults (tutorship or guardianship)
* fever ≥ 38.5°C
* chronic endstage kidney failure (Glomerular filtration rate < 30%)
* Solitary kidney
* Urinary tract catheter or percutaneous nephrectomy
* Pregnancy
* traumatic back pain
* Renal colic diagnosis in the past three months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2019-10-07 (Actual); Primary Completion 2020-07 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
Time between admission and discharge from the emergency room | Day one

SECONDARY OUTCOMES:
Patients satisfaction scale | An average of 24 hours
  5 questions to be answered by the patients rated on 1-10 scales being equivalent to 1 being equivalent to "no, certainly not and 10 being equivalent to "yes, certainly yes ". An overall score of 50 will be calculated to assess patient satisfaction.
Physician satisfaction scale | 9 months
  5 questions to be answered by the physicians rated on 1-10 scales being equivalent to 1 being equivalent to "no, certainly not and 10 being equivalent to "yes, certainly yes ". An overall score of 50 will be calculated to assess physician satisfaction.
Ultrasound diagnostic performance to detect expansions of the pelvicalyceal cavities | 9 months
  The diagnostic performance of the ultrasound for the detection of dilation of pyelocalicial cavities will be evaluated by sensitivity and specificity. The Gold Standard will be the result of the scanner

CONTACTS AND LOCATIONS:
Overall Officials: Duga Hervé, MD, Principal Investigator — GHICL
Locations (1):
- GHICL, Lille, France

IPD SHARING:
Plan to Share IPD: No